CLINICAL TRIAL: NCT03866109
Title: A Phase I/IIa Dose Escalation Study Evaluating the Safety and Efficacy of Autologous CD34+-Enriched HSPCs Genetically Modified With Human Interferon-α2 in Patients With Glioblastoma Multiforme and Unmethylated MGMT Gene Promoter
Brief Title: A Study Evaluating Temferon in Patients With Glioblastoma & Unmethylated MGMT
Acronym: TEM-GBM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genenta Science (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TEM-GBM_001; 2018-001404-11 (EudraCT Number); 2023-510299-29 (EudraCT Number)
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma Multiforme
Keywords: Temferon; Gene Therapy; Immunotherapy; Solid tumor
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Intervention Model Description: 8 cohorts: Cohorts 1-4, 6: Thiotepa and BCNU Conditioning; Temferon dose 0.5 - 3 x10^6 CD34+ cells/kg; Cohort 5: Thiotepa and Busulfan Condtioning; Temferon 2 x 10^6 CD34+ cells/kg; Cohort 7: Busulfan conditioning; Temferon 3 x 10^6 CD34+ cells/kg; Cohort 8: Busulfan conditioning; Temferon 4 x 10^6 CD34+ cells/kg;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temferon (Experimental): Autologous CD34+-enriched hematopoietic progenitor cells exposed in vitro to specific lentiviral vector encoding for the human interferon-alpha 2 gene. Its expression is tightly controlled by the human TIE2 enhancer/promoter sequence and by a post-transcriptional regulation layer represented by target miRNA sequences. This enables suppression of interferon-alpha2 expression in HSPCs, thereby further increasing the specificity of the delivery strategy for their Tie2 expressing myeloid cell progeny.
  Interventions: Drug: Temferon

INTERVENTIONS:
Drug: Temferon — Genetically modified HSPCs

SUMMARY:
This is a non-randomized, open label, phase I/IIa, dose-escalation study, involving a single injection of Temferon, an investigational advanced therapy consisting of autologous CD34+-enriched hematopoietic stem and progenitor cells exposed to transduction with a lentiviral vector driving myeloid specific interferon-alpha2 expression, which will be administered to up to 27 patients affected by GBM who have an unmethylated MGMT promoter. Part A will evaluate the safety and tolerability of 5 escalating doses of Temferon and 3 different conditioning regimens in up to 27 patients, following first line treatment.

DETAILED DESCRIPTION:
This is a non-randomized, open label, multicenter, phase I/IIa, therapeutic-exploratory, dose escalation, prospective study, involving a single injection of Temferon, an investigational ATMP consisting of autologous CD34+-enriched HSPCs exposed to transduction with a 3rd generation lentiviral vector driving myeloid-specific IFN-alpha2 expression, which will be administered to up to 27 patients affected by GBM who have an unmethylated MGMT promoter. The study will recruit and follow-up patients at a specialist neurosurgical and neuro-oncology units in Italy. Administration of Temferon and hematological follow up will take place at specialist hematology and bone marrow transplantation units.

Potentially eligible patients will be identified immediately after surgical resection of GBM once the MGMT promoter methylator status is known. Once written, informed consent is obtained, and screening procedures have been completed, harvesting of HSPCs will occur. A standard of care regimen lasting approximately 6 weeks, will then take place . During this time, Temferon manufacturing will occur. Following completion of radiotherapy, patients will be admitted for receipt of a conditioning regimen consisting of BCNU and thiotepa (Cohorts 1-6), busulfan and thiotepa (Cohort 5), or busulfan (Cohorts 7 and 8). This will be followed by administration of Temferon. In-patient monitoring will occur until hematological recovery occurs. Thereafter, regular follow-up of patients will occur up to 2 years (+720 days) with the majority of assessments and procedures. At the +720 day visit, patients will be invited to participate in a long term follow-up study which will last for an additional 6 years.

In Part A of the study, 8 cohorts of 3 patients will receive 5 escalating doses of Temferon. On completion of dose escalation in Part A, a conditioning regimen and single dose of Temferon will be selected to be studied in up to a further 6 patients.

In the event that GBM disease progression occurs, patients will be managed with second line therapies including second surgery, TMZ, BCNU, fotemustine or any other approved therapy for GBM.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed supratentorial glioblastoma with unmethylated MGMT gene promoter.
* Patients have undergone complete or partial tumor resection.
* Able and willing to provide written informed consent and comply with the study protocol and procedures.
* Eligible for radiotherapy.
* Life expectancy of 6 months or more at Screening.
* Women of child-bearing potential enrolled in the study must have a negative pregnancy test at screening and agree to use acceptable methods of contraception during the trial.
* Men enrolled in the study with partners who are women of child-bearing potential, must be willing to use an acceptable barrier contraceptive method during the trial or have undergone successful vasectomy at least 6 months prior to entry into the study. Successful vasectomy needs to have been confirmed by semen analysis.
* Karnofsky performance score (KPS)≥70.

Additional inclusion criteria to be assessed within 20 days of Temferon administration:

* Adequate cardiac, renal, hepatic and pulmonary function as evidenced by:
* Left ventricular ejection fraction (LVEF) ≥ 45% by echo and normal electrocardiogram (ECG) or presence of abnormalities not significant for cardiac disease.
* Absence of severe pulmonary hypertension;
* Diffusing capacity of the lung for carbon monoxide (DLCO) >50% and forced expiratory volume in 1 sec (FEV1) and forced expiratory vital capacity (FVC) > 60% predicted (if non cooperative: pulse oximetry > 95% in room air);
* Serum creatinine < 2x upper limit normal and estimated glomerular filtration rate (eGFR) ≥ 30ml/min/1.73m^2;
* Alkaline phosphatase (ALP), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 2.5 x upper limit of normal (ULN), and total bilirubin ≤ 2.0 mg/dl.
* Hemoglobin ≥10 g/dL, platelet count ≥100000/mm^3, absolute neutrophil count >1500/mm^3.

Exclusion Criteria:

* Use of other investigational agents or procedures within 4 weeks prior to study enrolment (within 6 weeks if use of long-acting agents) or participation in a previous gene therapy study.
* Known hypersensitivity to carmustine (or any other nitrosurea), busulfan, thiotepa, lenograstim, plerixafor, or any excipients used in these products.
* Receipt of any oral or parenteral chemotherapy or immunotherapy within 2 years of Screening.
* Previous allogeneic bone marrow transplantation, kidney or liver transplant.
* Clinical evidence of persistent raised intracranial pressure following surgical resection.
* Clinically relevant active viral, bacterial, or fungal infection at eligibility evaluation.
* Active autoimmune disease or a relevant history of important autoimmune manifestations, in particular psoriasis, systemic lupus erythematosus (SLE), rheumatoid arthritis, vasculitis, immunemediated peripheral neuropathies.
* History of sarcoidosis.
* History or current evidence of neuropsychiatric illness including depression, schizophrenia, bipolar disorders, impaired cognitive function, dementia or suicidal tendency.
* History of severe cardiovascular disease such as prior stroke, coronary artery disease requiring intervention or unresolved arrhythmias in the past 6 months.
* Evidence of any hematological neoplasm.
* Positivity for human immunodeficiency virus type 1 or 2 (HIV-1, HIV-2) (serology or RNA), and/or Hepatitis B Virus Surface Antigen (HbsAg) and/or Hepatitis B Virus (HBV) DNA and/or Hepatitis C virus (HCV) RNA (or negative HCV RNA but on antiviral treatment) and/or Treponema Pallidum or Mycoplasma active infection.
* Active alcohol or substance abuse within 6 months of the study.
* Current pregnancy or lactation.
* Known bleeding diathesis or history of abnormal bleeding, or any other known coagulation abnormalities that would contraindicate lumbar puncture for CSF or future surgery.
* Use of immunosuppressants with the exception of steroids. The maximum permitted dexamethasone (or equivalent) dose is 4 mg per day.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2019-03-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Tolerability and safety of Temferon over the first 90 days following administration as determined by the incidence of adverse events | 90 days
  Routine clinical and laboratory surveillance

SECONDARY OUTCOMES:
Long term tolerability and safety of Temferon as determined by the incidence of adverse events | 2 years
  Routine clinical and laboratory surveillance
Proportion of patients achieving haematologic recovery by Day +30 (defined as the first of at least 3 consecutive days with a neutrophil count >0.5 x 10^9/L and platelet count >20 x 10^9/L) | 30 days
  Hematologic recovery is defined as the first of at least 3 consecutive days with a neutrophil count >0.5 x 10^9/L and platelet count >20 x 10^9/L.
Determine the maximum tolerated dose of Temferon | 30 days
  Presence of a CTCAE Grade 3-5 adverse event (AE) that occurs within the first 30 days and is attributed to Temferon.
Identify presence of transduced myeloid cells in bone marrow as determined by vector copy number | Over 2 years
  VCN
Incidence of adverse events attributed to the conditioning regimen | Day +30
  Adverse events for BCNU and thiotepa, busulfan and thiotepa, or busulfan monotherapy up to Day +45
Identify presence of transduced myeloid cells in peripheral blood as determined by vector copy number | Over 2 years
  VCN
Determine clinical response in patients as determined by iRANO criteria | Over 2 years
  iRANO criteria
Determine progression free survival in patients | Over 2 years
  MRI
Determine overall survival in patients | 2 years
  Survival data
Changes in functional status (Eastern Cooperative Oncology Group) | 2 years
  ECOG assessment:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
Changes in functional status (Karnofsky) | 2 years
  Karnofsky assessment
Changes in Quality of Life (European Organisation for Research and Treatment of Cancer EORTC C30) | 2 years
  EORTC C30 questionnaire
Changes in Quality of Life (BN20) | 2 years
  European Organisation for Research and Treatment of Cancer BN20 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Finocchiaro, MD, Study Chair — Ospedale San Raffaele
Locations (3):
- Italy (3):
  - Ospedale San Raffaele, Milan
  - Fondazione IRCCS Istituto Neurologico "Carlo Besta", Milan
  - Policlinico Universitario Fondazione Agostino Gemelli, Rome

IPD SHARING:
Plan to Share IPD: No